CLINICAL TRIAL: NCT01254500
Title: To Investigate the Event Related Potentials (ERPs) of Patients With Brain Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sui Foon Lo, China Medical University Hospital
Other Study IDs: DMR-100-108
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Brain Lesions
Keywords: patients with brain lesions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- patients with brain lesions
- young normal controls
- old normal controls

SUMMARY:
Event-related potentials (ERPs）has the advantage of excellent temporal resolution on measuring real-time neural activities that reflect to higher level cognitive processes. A research project related to lesion studies in which patients with cognitive function impairment and communication disorder will be recruited as participants to examine their impairment as well as residual abilities by using ERPs. Hopefully, expected findings will provide further analysis based on the patterns of neural activities revealed by both patients and normal controls should be able to provide important evidence toward building the cross-linguistic theory. The findings also have applications on diagnostic and evaluation for patients with brain lesions for clinical application with communication disorder.

ELIGIBILITY:
Inclusion Criteria:

* patients with new brain lesions confirmed by imaging study

Exclusion Criteria:

* patients with recurrent brain lesions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with brain lesions young normal controls old normal controls
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan